CLINICAL TRIAL: NCT05120674
Title: The Nightmare Augmented Protocol for Treatment of Nightmares in Veterans With PTSD
Acronym: NAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study interrupted due to COVID-19 and then investigator changed institutions
Sponsor: VA Eastern Kansas (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christi M. Houston, PsyD, Principal Investigator, VA Eastern Kansas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH-0001
Record Dates: First submitted 2021-10-05; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPT+CBT-I (usual care) (Active Comparator): Veterans in this group completed the inpatient unit's existing Cognitive Processing Therapy (CPT) group based protocol. Furthermore, veterans in this group will also complete the inpatient unit's existing Cognitive Behavioral Therapy for Insomnia (CBT-I) group based protocol.
  Interventions: Behavioral: CPT; Behavioral: Cognitive Behavioral Therapy for Insomnia
- CPT+ CBT-I + ERRT (Active Comparator): Veterans in this group completed the CPT and CBT-I protocols augmented by the ERRT. ERRT therapy focuses on treating the posttrauma nightmares and does these via sleep hygiene, nightmare rescription, and exposure.
  Interventions: Behavioral: CPT; Behavioral: ERRT; Behavioral: Cognitive Behavioral Therapy for Insomnia
- CPT+ CBT-I + ERRT + NAP (Experimental): Veterans in this group will complete the CPT+CBT-I+ERRT protocol augmented by auditory stimulation (NAP). Exposure stimulation includes playing a rhythmic tone at 40-60hz (commonly referred to as pink noise) throughout the ERRT session and during the presleep exposure portion of ERRT. During the ERRT session, the tone will be played softly so as not to interfere with the session and will be played throughout the entire session. Before sleep, the veteran will play the 40-60hz tone via their smartphone while they read their rescripted nightmare. During sleep, the 40-60hz tone will be delivered during slow-wave-sleep (SWS) by the DREEM device (DREEM, 2013).
  Interventions: Behavioral: NAP; Behavioral: CPT; Behavioral: ERRT; Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: NAP — During the ERRT session, the tone will be played softly so as not to interfere with the session and will be played throughout the entire session. Before sleep, the veteran will play the 40-60hz tone via their smartphone while they read their rescripted nightmare. During sleep, the 40-60hz tone will be delivered during slow-wave-sleep (SWS) by the DREEM device. The pairing of the tone with the intervention is expected to trigger benefits of the exercise in reducing nightmare disturbance during sleep.
  Arms: CPT+ CBT-I + ERRT + NAP
Behavioral: CPT — Cognitive Therapy for PTSD
  Other Names: Cognitive Processing Therapy
Behavioral: ERRT — ERRT asks individuals to rewrite the traumatic event that triggered their nightmares and then review the rescription before bed. This technique has been proven to drastically reduce the frequency of chronic nightmares.
  Other Names: Exposure, Relaxation, and Rescripting Therapy
  Arms: CPT+ CBT-I + ERRT; CPT+ CBT-I + ERRT + NAP
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia that includes behavioral and cognitive interventions related to sleep hygiene, increasing sleep drive, and modifying behaviors that result in association between laying in bed and wakeful states.
  Other Names: CBT-I

SUMMARY:
The primary goal of this study is to determine whether the use of a timed tone played during sleep, in addition to the use of established therapies, will reduce or eliminate the occurrence of nightmares. In particular, the protocol tests two different mechanisms for improvement: 1) further decreasing autonomic arousal and providing a mechanism for restoration and 2) enhancing memory processing for the alternate version of the traumatic events.

DETAILED DESCRIPTION:
Study Population: The study population consisted of veterans who experienced nightmares and were enrolled in a voluntary inpatient stress unit at the Topeka VA. Given that individuals enrolled in the inpatient unit were under constant treatment conditions, there are no specific demographic requirements for this study.

Participants were informed about the study and, if interested, completed the informed consent process. Consented participants were randomly assigned to a treatment group. Self-reported symptoms (e.g., sleep duration, quality, presence and severity of nightmares) were assessed every morning via sleep diaries and sleep was recorded objectively via the DREEM device. Participants were debriefed upon completion of treatment.

All participants who consent for participation and meet inclusion/exclusion criteria were randomly assigned into one of three potential groups. Participants were randomly sorted into groups via an ordered systematic separation pattern. Both participants and data analysts were blinded to the group assignments. Specific protocol details for each group are described below. Regardless of group assignment, all participants followed the treatment unit's standard protocols, with the only change being that Groups 2 (Cognitive Processing Therapy + Cognitive Behavioral Therapy for Insomnia) & 3 (Cognitive Processing Therapy + Cognitive Behavioral Therapy for Insomnia + Nightmare Augmented Protocol-NAP) participated in an Exposure, Relaxation, and Rescripting Therapy (ERRT) and Group 1 (Cognitive Processing Therapy only group) did not.

The NAP intervention: Veterans in group 3 completed the Cognitive Processing Therapy +ERRT protocol augmented by the auditory stimulation delivered by the DREEM device. Auditory stimulation consists of exposure and sleep stimulation. Exposure stimulation includes playing a rhythmic tone at 40-60hz (commonly referred to as pink noise) throughout the ERRT session and during the presleep exposure portion of ERRT. During the ERRT session, the tone will be played softly so as not to interfere with the session and will be played throughout the entire session. Before sleep, the veteran played the 40-60hz tone via their smartphone while they read their rescripted nightmare. During sleep, the 40-60hz tone was delivered during slow-wave-sleep (SWS) by the DREEM device. The DREEM device is a headband like device used to measure and enhance sleep via auditory stimulation. The DREEM device uses electroencephalogram (EEG) to determine when an individual is in SWS and then uses built in speakers to play the desired tone (this tone is undetectable to the dreamer and will not wake them). The DREEM device has been demonstrated to be a safe and effective device for measuring and enhancing sleep.

Data Collection: Presleep arousal, sleep quality, and the occurrence of a posttrauma nightmare(s) were assessed via sleep diaries. Sleep diaries were completed every night prior to bedtime and every morning upon awakening. Each daily diary consisted of outcome measures including the Nightmare Diary entry, Presleep Arousal Scale (PAS), Morning Diary entry, Pittsburgh Sleep Quality Index (PSQI), and the Trauma-Related Nightmare Survey (TRNS).

Statistical Analyses: Repeated measures Analysis of Variance (ANOVA) will be used to compare nightmare frequency and sleep quality both within and between treatment groups. These analyses will be used to determine if groups had significant reductions in nightmare frequency/ improvements in sleep quality improvement and to determine if there are group differences in sleep quality. For participants in the NAP group, the researchers will use multilevel modeling (MLM) to determine whether there were changes in sleep macro or micro architecture concurrent with introduction of the auditory tone.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans enrolled in the inpatient stress unit.
2. Veterans who consent to participating in the treatment study.
3. Veterans who report experiencing weekly nightmares related to a traumatic event.

Exclusion Criteria:

1. Does not own a smartphone that can access the internet.
2. Veterans who do not experience nightmares related to a traumatic event.
3. Veterans who are unable to wear an electronic headband during sleep.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | through study completion, an average of 1 month
  The PSQI is a self-report measure designed to assess certain qualities and problems associated with sleep. Participants rate quality of sleep and degree of sleep difficulties for the month preceding the assessment. A global sleep quality score is obtained by summing the seven component scores including: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Higher scores reflect poorer sleep quality. The global score ranges from 0-21. A cut-off score of 5 as distinguishing "good" sleepers from "poor" sleepers with a diagnostic sensitivity of 89.6% and specificity of 86.5%. The PSQI was adapted for daily usage following standard protocols.
Trauma-Related Nightmare Survey (TRNS) | through study completion, an average of 1 month
  The TRNS is a self-report measure developed for the assessment of nightmares and related sleep disturbance. The TRNS was adapted for daily usage following standard protocols.

SECONDARY OUTCOMES:
Presleep Arousal Scale (PAS) | through study completion, an average of 1 month
  The PAS is a self-report measure designed to assess somatic and cognitive arousal prior to sleep. Furthermore, the PAS can be combined to assess overall presleep arousal. The PAS has been found to be a reliable and valid measure of arousal. Cronbach's αs of the Cognitive and Somatic subscales were, respectively, 0.88 and 0.79. Furthermore, all item-subscale correlations are highly significant and in the predicted direction (all rs significant at p < 0.01). The PAS was updated for daily use.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Eastern Kansas, Leavenworth, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT05120674/ICF_000.pdf